CLINICAL TRIAL: NCT02443467
Title: A Study to Determine the Safety and Tolerability of Herceptin as an Adjuvant Therapy of Early Breast Cancer
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML20397
Record Dates: First submitted 2015-05-11; First posted 2015-05-13 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Breast Cancer, Early Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- HER2-positive early breast cancer: Human Epidermal Growth Factor Receptor 2 (HER2)-positive early breast cancer treated with loading dose of Herceptin (trastuzumab) administered as 6 mg/kg followed by once in 3 weeks administration at 4 mg/kg up to 12 months of treatment
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
This was an open-labeled, multi-center, prospective, non-comparative study of the safety of Herceptin (trastuzumab) used as an adjuvant therapy in patients with early breast cancer who had previously received antracycline therapy before or after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Female patients > or = 18 years of age
* Human Epidermal Growth Factor Receptor 2 (HER2)-neu overexpression
* Previously treated with adjuvant antracycline containing chemotherapy
* Left Ventricular Ejection Fraction (LVEF) > 50%
* Eastern Cooperative Oncology Group (ECOG) score < or = 2
* Life expectancy > or = 12 weeks

Exclusion Criteria:

* Left Ventricular Ejection Fraction (LVEF) < 50%
* Advanced pulmonary disease
* Severe dyspnea
* Abnormal laboratory results within 14 days prior to registration
* Peripheral neuropathy
* Presence of Central Nervous System (CNS) metastasis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with HER2-positive early breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2006-07; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with adverse events | Up to 3 years
Percentage of participants with serious adverse events | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Kamenitz, Serbia